CLINICAL TRIAL: NCT00985985
Title: A Multi-center, Randomized, Double-blind, Parallel, Placebo-controlled Clinical Study to Evaluate Efficacy and Safety of Nicotine Mint Lozenge (2mg and 4mg) in Smoking Cessation
Brief Title: Efficacy and Safety Study of Nicotine Mint Lozenge (2mg and 4mg) in Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHN-Nicotine Mint Lozenge-002
Record Dates: First submitted 2009-09-02; First posted 2009-09-29 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Smoking
Keywords: smoking cessation; nicotine lozenge; nicotine replacement therapy
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2mg nicotine lozenge (Experimental): 2 mg nicotine lozenge
  Interventions: Drug: Nicotine
- 2 mg placebo (Placebo Comparator): 2 mg placebo
  Interventions: Drug: Placebo
- 4 mg nicotine lozenge (Experimental): 4 mg nicotine lozenge
  Interventions: Drug: Nicotine
- 4 mg placebo (Placebo Comparator): 4 mg placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotine — 2 mg or 4 mg nicotine lozenge
  Arms: 2mg nicotine lozenge; 4 mg nicotine lozenge
Drug: Placebo — placebo lozenge
  Arms: 2 mg placebo; 4 mg placebo

SUMMARY:
A multi-center, randomized, double-blind, placebo-controlled, 4-arm clinical study to evaluate efficacy and safety of nicotine lozenge (2mg and 4mg) in smoking cessation in adult cigarette smokers who are motivated to quit smoking. Successful quitters or participants who smoke occasionally will be followed up after week 24 till 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age or older;
* Participant is motivated in smoking cessation using nicotine mint lozenge;
* Participant has the habit of smoking regularly every day for at least 1 year;
* Participant is able to read and provide written informed consent.

Exclusion Criteria:

* Participant uses other forms of tobacco other than cigarettes such as pipes, cigars, snuff, or smokeless tobacco within 30 days of entry into the study;
* Participant uses other nicotine delivery system such as nicotine gum, nicotine patch, nicotine inhaler, or nicotine nasal spray etc. within 30 days of study entry;
* Participant smoke any other substance within 30 days of study entry (such as cannabis, cocaine, heroin, ice drug, herbal cigarettes etc);
* The participant has a past history of alcohol or drug abuse;
* Participants use other smoking cessation aids (including bupropion, varenicline, traditional Chinese medicines such as herbals, acupuncture, consultation etc), within 30 days of study entry.;
* Participant is currently involved in another clinical trial or has used any investigational medication within 30 days of study entry; Any previous participation in this study;
* Participant is a member of the same household as another clinical subject. Subject is a relative of study site staff or member of the study staff;
* Participant is pregnant or breast-feeding, or has childbearing potential but refusing taking medical contraception measures (within first 24 weeks during study). (Note: All female subjects with childbearing potential must take urine pregnancy test before entry the study, only negative result subject is permitted to this study.);
* Participants who have heart and cerebral vascular disease not stable or controlled by medication or have an irregular heartbeat or have had a heart attack within the last 3 months;
* Participants with poorly controlled high blood pressure by medications, systolic BP greater than or equal to 140mmHg, diastolic BP greater than or equal to 90mmHg after administration;
* Participants having hyperthyroidism or current application of insulin for diabetes;
* Participants having myocardial infarction or cerebral vascular accidents recently (within the past 3 months);
* Participants who are unable to fulfill study requirements in relation to conforming to the visit schedule;
* Participants who are allergy to Aspartame or Phenylpyruvic acid (an edulcorant is widely used in foods and drinks)，or have diagnosed with Phenylketonuria;
* The other clinically significant pulmonary, gastrointestinal, liver, neurological, renal or haematological abnormalities.( unstable or worsening angina pectoris, Prinzmetal's angina, nerve or circulatory problems, rheumatoid arthritis, moderate and severe COPD);
* A medical history that, in the opinion of the investigator, might jeopardize the safety of the subject or the validity for the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 723 (Actual)
Dates: Start 2009-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Of 781 screened participants, only 723 were randomized and remaining 58 were considered screening failures. Participants who smoked their first cigarette within 30 minutes after waking were considered as high dependence smokers while those who smoked their first cigarette after 30 minutes of waking were considered as low dependence smokers.
Groups:
- Nicotine Lozenge 2 Milligram (mg) (Low Dependence Smokers): Participants who smoked their first cigarette after 30 minutes of waking received 2 mg of nicotine lozenge, orally. During week 1 to week 6,participants were recommended to take at least 9 lozenges per day, but not exceeding 15 lozenges. During week 7 to week 9, participants were recommended to use 12 to 6 lozenges per day, further taking 3 to 6 lozenges only by week 10 to 12. Afterwards, lozenge was taken when necessary to prevent relapse.
- Placebo Lozenge (Low Dependence Smokers): Participants who smoked their first cigarette after 30 minutes of waking received placebo lozenge containing 0 mg of nicotine, orally. During week 1 to week 6, participants were recommended to take atleast 9 lozenges per day but not exceeding 15 lozenges. During week 7 to week 9, participants were recommended to use 12 to 6 lozenges per day, further taking 3 to 6 lozenges only by week 10 to 12. Afterwards, lozenge was taken when necessary to prevent relapse
- Nicotine Lozenge 4 mg (High Dependence Smokers): Participants who smoked their first cigarette within 30 minutes after waking received 4 mg nicotine lozenge, orally. During week 1 to week 6, participants were recommended to take at least 9 lozenges per day but not exceeding 15 lozenges. During week 7 to week 9, participants were recommended to use 12 to 6 lozenge per day, further taking 3 to 6 lozenges only by week 10 to 12. Afterwards, lozenge was taken when necessary to prevent relapse.
- Placebo Lozenge (High Dependence Smoke: Participants who smoked their first cigarette within 30 minutes after waking received placebo lozenge containing 0 mg of nicotine, orally. During week 1 to week 6, participants were recommended to take at least 9 lozenges per day but not exceeding 15 lozenges. During week 7 to week 9, participants were recommended to use 12 to 6 lozenge per day, further taking 3 to 6 lozenges only by week 10 to 12. Afterwards, lozenge was taken when necessary to prevent relapse.
Period: Overall Study
Arm/Group | Nicotine Lozenge 2 Milligram (mg) (Low Dependence Smokers) | Placebo Lozenge (Low Dependence Smokers) | Nicotine Lozenge 4 mg (High Dependence Smokers) | Placebo Lozenge (High Dependence Smoke
Started | 241 | 242 | 120 | 120
Safety Population | 241 | 242 | 119 | 118
Full Analysis Set (FAS) Population | 241 | 242 | 120 | 119 (One participant withdrew consent and was not included as the FAS population.)
Completed | 217 | 218 | 109 | 107
Not Completed | 24 | 24 | 11 | 13
Not completed — Adverse Event | 4 | 2 | 2 | 2
Not completed — Lost to Follow-up | 4 | 11 | 2 | 3
Not completed — Protocol Violation | 1 | 2 | 0 | 1
Not completed — Lack of Efficacy | 5 | 6 | 1 | 3
Not completed — Withdrawal by Subject | 4 | 2 | 2 | 2
Not completed — Other Reason | 6 | 1 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Nicotine Lozenge 2 mg (Low Dependence Smokers): Participants who smoked their first cigarette after 30 minutes of waking received 2 mg of nicotine lozenge, orally.
- Placebo Lozenge (Low Dependence Smokers): Participants who smoked their first cigarette after 30 minutes of waking received placebo lozenge containing 0 mg of nicotine, orally.
- Nicotine Lozenge 4 mg (High Dependence Smokers): Participants who smoked their first cigarette within 30 minutes after waking received 4 mg nicotine lozenge, orally.
- Placebo Lozenge (High Dependence Smokers): Participants who smoked their first cigarette within 30 minutes after waking received placebo lozenge containing 0 mg of nicotine, orally.
- Total: Total of all reporting groups
Arm/Group | Nicotine Lozenge 2 mg (Low Dependence Smokers) | Placebo Lozenge (Low Dependence Smokers) | Nicotine Lozenge 4 mg (High Dependence Smokers) | Placebo Lozenge (High Dependence Smokers) | Total
Number analyzed (Participants) | 241 | 242 | 120 | 119 | 722
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline parameters were evaluated for FAS population.
  Years | 38.4 (11.78) | 39.9 (11.76) | 42.3 (10.38) | 42.0 (10.57) | 40.1 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline parameter were evaluated for FAS population.
  Participants
    Female | 11 | 7 | 2 | 3 | 23
    Male | 230 | 235 | 118 | 116 | 699
Body Weight [Mean (Standard Deviation); unit: Kg] — Baseline Parameters were evaluated for FAS population.
  Kg | 71.8 (11.06) | 72.3 (11.42) | 75.9 (11.64) | 74.3 (12.15) | 73.1 (11.53)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Successful Smoking Cessation at Week 6
Description: Rate of Successful Smoking Cessation at Week 6 was measured by Carbon Monoxide (CO) breath levels.
Time Frame: From baseline to Week 6
Population: Analysis was considered per Full Analysis Set (FAS) population. FAS population consisted of all randomized participants who had study medication for at least once with assessment data post-dosing.
Measure: Number; unit: Percentage of participants
Groups:
- Nicotine Lozenge 2 mg (Low Dependence Smokers): Participants, who smoked their first cigarette after 30 minutes of waking, received 2 mg of nicotine lozenge orally.
- Placebo Lozenge (Low Dependence Smokers): Participants, who smoked their first cigarette after 30 minutes of waking, received placebo lozenge containing 0 mg of nicotine orally.
- Nicotine Lozenge 4 mg (High Dependence Smokers): Participants, who smoked their first cigarette within 30 minutes after waking, received 4 mg nicotine lozenge orally.
- Placebo Lozenge (High Dependence Smokers): Participants, who smoked their first cigarette within 30 minutes after waking, received placebo lozenge containing 0 mg of nicotine orally.
Arm/Group | Nicotine Lozenge 2 mg (Low Dependence Smokers) | Placebo Lozenge (Low Dependence Smokers) | Nicotine Lozenge 4 mg (High Dependence Smokers) | Placebo Lozenge (High Dependence Smokers)
Number analyzed (Participants) | 241 | 242 | 120 | 119
Percentage of participants | 24.48 | 21.49 | 30.83 | 20.17
Statistical Analysis 1: Comparison: Nicotine Lozenge 2 mg (Low Dependence Smokers) vs Placebo Lozenge (Low Dependence Smokers); Null hypothesis considered no treatment difference in the smoking cessation success rate for the active treatment versus its matching placebo; Test type: Superiority or Other; p = 0.3851, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.78 to 1.92] — Odds Ratio based on logistic model (adjusted by center)
Statistical Analysis 2: Comparison: Nicotine Lozenge 4 mg (High Dependence Smokers) vs Placebo Lozenge (High Dependence Smokers); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0565, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.99 to 3.32] — Odds Ratio based on logistic model (adjusted by center)

2. Secondary Outcome: Rate of Continuous Successful Smoking Cessation at Week 12 and Week 24
Description: Continuous abstinence was verified by measurement of CO breath levels.
Time Frame: From baseline to Week 12 and Week 24
Population: Analysis was done per FAS population. FAS population consisted of all randomized subjects who had study medication for at least once with assessment data post-dosing.
Measure: Number; unit: Percentage of participants
Arm/Group | Nicotine Lozenge 2 mg (Low Dependence Smokers) | Placebo Lozenge (Low Dependence Smokers) | Nicotine Lozenge 4 mg (High Dependence Smokers) | Placebo Lozenge (High Dependence Smokers)
Number analyzed (Participants) | 241 | 242 | 120 | 119
Percentage of participants
  Smoking Cessation Rate at 12 weeks | 17.84 | 16.94 | 22.50 | 10.92
  Smoking Cessation Rate at 24 weeks | 12.86 | 13.22 | 19.17 | 10.08

3. Secondary Outcome: Rate of Long-term Successful Smoking Cessation at Week 24
Description: Rate of long-term successful smoking cessation at Week 24 was defined as the proportion of participants who achieved the primary end-point with no more than six cumulative days of smoking from Week 6 to Week 24.
Time Frame: From Week 6 to Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Nicotine Lozenge 2 mg (Low Dependence Smokers) | Placebo Lozenge (Low Dependence Smokers) | Nicotine Lozenge 4 mg (High Dependence Smokers) | Placebo Lozenge (High Dependence Smokers)
Number analyzed (Participants) | 241 | 242 | 120 | 119
Percentage of participants | 19.09 | 17.77 | 24.17 | 15.97

4. Secondary Outcome: Proportion of Participants With Seven Day Point Prevalence Abstinence
Description: Seven day point prevalence abstinence was defined as complete abstinence from smoking for the 7 days up to and including the evaluation day.
Time Frame: Weekly assessment at Week 1, 2, 4, 6, 12 and Week 24
Population: Analysis was carried out per FAS population. FAS population consisted of all randomized subjects who had study medication for at least once with assessment data post-dosing.
Measure: Number; unit: Percentage of participants
Arm/Group | Nicotine Lozenge 2 mg (Low Dependence Smokers) | Placebo Lozenge (Low Dependence Smokers) | Nicotine Lozenge 4 mg (High Dependence Smokers) | Placebo Lozenge (High Dependence Smokers)
Number analyzed (Participants) | 241 | 242 | 120 | 119
Percentage of participants
  Week 1 | 12.45 | 11.98 | 20.00 | 10.08
  Week 2 | 21.16 | 23.14 | 33.33 | 26.05
  Week 4 | 31.95 | 29.34 | 36.67 | 30.25
  Week 6 | 35.68 | 37.19 | 41.67 | 32.77
  Week 12 | 41.49 | 39.26 | 40.83 | 26.05
  Week 24 | 41.49 | 43.80 | 50.00 | 43.70

5. Secondary Outcome: Mean Score of Relief of Craving/ Total Withdrawal Symptoms
Description: The evaluation of withdrawal and craving symptoms was carried out every day with the Minnesota Nicotine Withdrawal scale (MNWS). The MNWS total score contains 9 items (urge to smoke; depressed mood; irritability, frustration, or anger; anxiety; difficulty concentrating; restlessness; increased appetite; difficulty going to sleep; difficulty staying asleep). Each item was rated on a 5 grade scale with scores ranging from 0 (best score) to 4 (worst score) i.e. none (score=0), slight (score=1), mild (score=2), moderate (score=3), and severe (score=4). For each symptom at each week, the average score was calculated as the average of the daily scores during that week. The total score was calculated as the sum of the 9 symptoms.
Time Frame: Weekly assessment at Week 1, 2, 3, 4, 5 and Week 6
Population: Analysis was carried out per FAS population, which consisted of all randomized subjects who have had study medication for at least once with assessment data post-dosing. Due to drop outs, there was difference in the number of participants analyzed (n) for this outcome measure. Missing values were not imputed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Placebo Lozenge (High Dependence Smokers): Participants, who smoked their first cigarette within 30 minutes after waking, received placebo lozenge containing 0 mg of nicotine, orally.
Arm/Group | Nicotine Lozenge 2 mg (Low Dependence Smokers) | Placebo Lozenge (Low Dependence Smokers) | Nicotine Lozenge 4 mg (High Dependence Smokers) | Placebo Lozenge (High Dependence Smokers)
Number analyzed (Participants) | 236 | 238 | 119 | 118
Score on a scale
  Week 1 (n=236, 238, 119, 118) | 8.40 (7.18) | 7.77 (6.55) | 7.66 (6.08) | 8.67 (7.02)
  Week 2 (n=230, 233, 112, 115) | 7.59 (7.25) | 6.84 (6.05) | 6.70 (5.96) | 7.39 (6.12)
  Week 3 (n=226, 232, 115, 110) | 6.80 (7.12) | 6.06 (5.83) | 6.17 (6.40) | 6.90 (5.97)
  Week 4 (n=225, 226, 113, 108) | 6.67 (7.36) | 5.45 (5.59) | 5.66 (6.19) | 6.71 (6.06)
  Week 5 (n=221, 229, 112, 104) | 6.06 (6.57) | 5.29 (5.72) | 5.60 (5.98) | 6.60 (5.94)
  Week 6 (215, 223, 103, 102) | 5.85 (6.53) | 5.45 (6.02) | 5.21 (5.58) | 6.49 (6.23)

6. Secondary Outcome: Mean Daily Dose at Visit 4, 5, 6, 7 and 10
Description: Mean daily dose of lozenges was calculated as number of lozenges taken at each visit divided by days since the last visit.
Time Frame: Weeks 1-2, 3-4, 5-6, 7-12 and 13-24
Population: Analysis was carried out per FAS population, which consisted of all randomized subjects who had study medication for at least once with assessment data post-dosing. Due to drop outs, there was difference in the population analyzed (n) for this outcome measure at each time point. Missing values were not imputed.
Measure: Mean (Standard Deviation); unit: Number of lozenges
Arm/Group | Nicotine Lozenge 2 mg (Low Dependence Smokers) | Placebo Lozenge (Low Dependence Smokers) | Nicotine Lozenge 4 mg (High Dependence Smokers) | Placebo Lozenge (High Dependence Smokers)
Number analyzed (Participants) | 232 | 237 | 117 | 111
Number of lozenges
  Week 1-2 (n=232, 237, 117, 111) | 8.96 (3.32) | 8.59 (3.23) | 8.81 (3.57) | 8.52 (3.16)
  Week 3-4 (n=224, 231, 114, 107) | 8.66 (3.17) | 8.71 (3.40) | 8.93 (3.17) | 8.60 (3.39)
  Week 5-6 (n=223, 228, 113, 106) | 8.15 (3.39) | 8.07 (3.30) | 8.55 (3.32) | 8.09 (3.43)
  Weeks 7-12 (n=221, 224, 112, 106) | 4.85 (2.33) | 4.54 (2.40) | 5.02 (2.35) | 4.67 (2.31)
  Weeks 13-24 (n=222, 222, 105, 107) | 0.89 (1.05) | 0.78 (1.04) | 0.95 (0.90) | 0.84 (0.92)

7. Secondary Outcome: Mean Change From Baseline in Body Weight at Week 6, Week 12 and Week 24/ Premature Termination.
Description: Change in body weight was analyzed at Weeks 6, 12, and 24.
Time Frame: Baseline, Week 6, 12 and Week 24
Population: Analysis was carried out per FAS population, which consisted of all randomized subjects who had study medication for at least once with assessment data post-dosing. Due to drop outs, there was difference in the population analyzed (n) for this outcome measure at each time point i.e. Week 6, Week 12 and Week 24. Missing values were not imputed.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Groups:
- Nicotine Lozenge 2 mg (Low Dependence Smokers): Participants, who smoked their first cigarette after 30 minutes of waking, received 2 mg of nicotine lozenge, orally.
Arm/Group | Nicotine Lozenge 2 mg (Low Dependence Smokers) | Placebo Lozenge (Low Dependence Smokers) | Nicotine Lozenge 4 mg (High Dependence Smokers) | Placebo Lozenge (High Dependence Smokers)
Number analyzed (Participants) | 241 | 242 | 120 | 119
kilogram (kg)
  Week 6 (n=225, 230, 115, 109) | 0.9 (1.94) | 0.7 (2.21) | 1.2 (2.45) | 1.2 (2.16)
  Week 12 (n=221, 225, 112, 107) | 1.2 (2.43) | 1.0 (2.40) | 1.9 (3.58) | 1.5 (2.17)
  Week 24 (n=221, 224, 111, 112) | 1.3 (2.89) | 1.3 (2.81) | 2.2 (3.14) | 2.1 (2.50)

8. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Cardiovascular AEs and Who Discontinued Due to AEs
Description: All AEs and SAEs were reviewed and reported by investigator. AEs were graded on a 3-point scale as Mild, Moderate and Severe.
Time Frame: Weekly assessments from first treatment dose up to 15 days after last treatment dose
Population: Safety Population of this study consists of all randomized participants who have had study medication for at least once.
Measure: Number; unit: Participants
Groups:
- Placebo Lozenge (Low Dependence Smokers): Participants, who smoked their first cigarette after 30 minutes of waking, received placebo lozenge containing 0 mg of nicotine, orally.
- Nicotine Lozenge 4 mg (High Dependence Smokers): Participants, who smoked their first cigarette within 30 minutes after waking received 4 mg nicotine lozenge, orally.
- Placebo Lozenge (High Dependence Smokers): Participants, who smoked their first cigarette within 30 minutes after waking received placebo lozenge containing 0 mg of nicotine, orally.
Arm/Group | Nicotine Lozenge 2 mg (Low Dependence Smokers) | Placebo Lozenge (Low Dependence Smokers) | Nicotine Lozenge 4 mg (High Dependence Smokers) | Placebo Lozenge (High Dependence Smokers)
Number analyzed (Participants) | 241 | 242 | 119 | 118
Participants
  AEs | 111 | 91 | 61 | 58
  SAEs | 1 | 0 | 1 | 1
  Cardiovascular AEs | 24 | 3 | 11 | 10
  Discontinuation due to AEs | 3 | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: All adverse events that occured in time-period from the first administration of product to up to 15 days after the last dosing were recorded
Description: Safety evaluation was done for saftey set population. There was one additional subject, randomized to 4mg Placebo, who withdrew consent, but was excluded from the SS population.
Groups:
- Nicotine Lozenge 2 mg (Low Dependence Smokers): Participants who smoked their first cigarette after 30 minutes after waking received 2 mg of nicotine lozenge, orally.
- Placebo Lozenge (Low Dependence Smokers): Participants who smoked their first cigarette after 30 minutes after waking received placebo lozenge containing 0 mg of nicotine, orally.
- Nicotine Lozenge 4 mg (High Dependence Smokers): Participants who smoked their first cigarette within 30 minutes after waking received 4 mg of nicotine lozenge, orally.
Arm/Group | Nicotine Lozenge 2 mg (Low Dependence Smokers) | Placebo Lozenge (Low Dependence Smokers) | Nicotine Lozenge 4 mg (High Dependence Smokers) | Placebo Lozenge (High Dependence Smokers)
Serious Adverse Events (participants affected / at risk) | 1/241 | 0/242 | 1/119 | 1/118
Other Adverse Events (participants affected / at risk) | 59/241 | 45/242 | 43/119 | 26/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Lozenge 2 mg (Low Dependence Smokers) (N=241) | Placebo Lozenge (Low Dependence Smokers) (N=242) | Nicotine Lozenge 4 mg (High Dependence Smokers) (N=119) | Placebo Lozenge (High Dependence Smokers) (N=118)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotine Lozenge 2 mg (Low Dependence Smokers) (N=241) | Placebo Lozenge (Low Dependence Smokers) (N=242) | Nicotine Lozenge 4 mg (High Dependence Smokers) (N=119) | Placebo Lozenge (High Dependence Smokers) (N=118)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 16 | 14 | 13 | 5
Nausea (Gastrointestinal disorders) | 15 | 10 | 7 | 8
Dyspnoea (Cardiac disorders) | 1 | 2 | 6 | 2
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 27 | 19 | 17 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.